CLINICAL TRIAL: NCT00150189
Title: Efficacy of Oral Sucrose Analgesia During Routine Immunizations at 6 Weeks and 4 Months of Age
Brief Title: Utilization of Oral Sucrose to Decrease Pain in Infants During Immunizations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB NO. 2003-315
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2006-12

CONDITIONS: Pain; Procedural Pain
Keywords: Pain; Procedural Pain; Sucrose; Infant; Newborn
MeSH Terms: conditions — Pain; Pain, Procedural | interventions — Sucrose

INTERVENTIONS:
Behavioral: Sucrose

SUMMARY:
The study explores the potential benefits of a sugar water solution for decreasing pain in infants during routine immunizations.

DETAILED DESCRIPTION:
Acute pain during early life may alter infant pain responses, cognitive development, and behavioral outcomes. Immunization injections represent a relatively brief exposure to acute pain, yet assessment studies demonstrate that infants respond with significant distress during the injections. This study will examine the analgesic potential of oral sucrose in diminishing the pain associated with immunization injections in 6 week to 4-month-old infants. The proposed mechanism of action is via the activation of endogenous opioids that attenuate nociceptive information at the level of the dorsal horn.

Comparison: Administration of oral sucrose 2 minutes prior to immunizations compared to administration of sterile water 2 minutes prior to immunizations

ELIGIBILITY:
Inclusion Criteria:

* Currently between 2 and 4 months of age
* Birth between 37 and 42 weeks' completed gestation;
* Birth weight greater than 2.5 kg
* No evidence of acute or chronic disease processes.

Exclusion Criteria:

* They are experiencing concurrent illness
* They received an analgesic/sedative 6 hours prior to the office visit
* The infant has breast fed 30 minutes prior to the visit or wishes to breast feed during or immediately after the immunization
* The infant has been introduced to solid food
* The infant may not receive a pacifier
* The infant is diagnosed with a major congenital disorder where the behavioral responses to painful stimuli may be altered
* Language barriers preclude the process of obtaining parental consent.

Ages: 6 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140
Dates: Start 2003-11-01 (Actual); Primary Completion 2006-10-11 (Actual); Study Completion 2006-10-11 (Actual)

PRIMARY OUTCOMES:
The University of Wisconsin Children's Hospital Pain Scale will measure the primary outcome acute behavioral pain response. Measure will be recorded at baseline, immediately after immunizations and 3 minutes following immunizations

SECONDARY OUTCOMES:
Duration of analgesia during immunizations
Age related changes in behavioral pain response during immunizations

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Hatfield, PhD(c) CNNP, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center'
Locations (1):
- General Ambulatory Pediatric Clinic, Penn State Children's Hospital, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Hatfield LA, Gusic ME, Dyer AM, Polomano RC. Analgesic properties of oral sucrose during routine immunizations at 2 and 4 months of age. Pediatrics. 2008 Feb;121(2):e327-34. doi: 10.1542/peds.2006-3719. PMID 18245406